CLINICAL TRIAL: NCT07008209
Title: Comparing the Effects of Reconstrual and Repurposing Reappraisal Strategies on Sadness and Anxiety in Emerging Adults: A Brief Intervention
Brief Title: Comparing the Effectiveness of Reappraisal Strategies in Adult Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Meryem Söğüt Kahramanlar, PhD(c), Ibn Haldun University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: E-71395021-050.04-50851
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Emotional Dysregulation; Anxiety; Sadness; Anxiety Disorders and Symptoms; Depressive Symptoms
Keywords: emotion regulation; reappraisal; cognitive reappraisal; repurposing; reconstrual; anxiety; sadness; emerging adults
MeSH Terms: conditions — Anxiety Disorders; Depression; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study uses a 2 (Emotion Type: Sadness vs. Anxiety) × 4 (Strategy Type: Reconstrual, Repurposing, Active Control, Passive Control) between-subjects factorial design. Participants are randomly assigned to one of eight experimental groups. Each participant is exposed to an emotionally evocative scenario (either sadness or anxiety), followed by an intervention based on their assigned strategy condition. The aim is to examine the main and interaction effects of strategy type and emotion type on changes in emotional experience before and after the intervention.
  Study Type: Interventional Design: Randomized, 2 × 4 between-subject factorial design Factors: Emotion Type (Sadness vs. Anxiety) × Strategy (Reconstrual, Repurposing, Active Control, Passive Control) Within-Subjects: Time (Post-Scenario vs. Post-Intervention) Allocation: Randomized Masking: Single-blind Primary Purpose: Basic Science
Who Masked: Investigator
Masking Description: This study uses an online platform (Qualtrics) to assign participants randomly to study arms and deliver interventions. Investigators are blinded to group allocation. Investigators do not have access to or control over assignment information during data collection, ensuring masking (single-blind design).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Sadness - Reconstrual (Experimental): Participants in this arm are exposed to sadness-related scenario and trained to use the reconstrual strategy, which involves reinterpreting the meaning of the situation to reduce negative emotions. Training is delivered online via Qualtrics and includes practice vignette. After training, participants apply reconstrual to the scenario to regulate their emotional response.
  Interventions: Behavioral: Reconstrual Strategy Training
- Sadness - Repurposing (Experimental): Participants view sadness-related scenario and receive training in repurposing, which focuses on changing the goal to alleviate negative feelings. Training and practice exercises are provided online through Qualtrics before applying the strategy to the scenario.
  Interventions: Behavioral: Repurposing Strategy Training
- Sadness - Active Control (Active Comparator): Participants are presented with sadness-related scenario followed by a writing distraction task designed to divert attention from negative emotions. This arm controls for the effect of engaging in an active cognitive task unrelated to emotion regulation.
  Interventions: Behavioral: Active Control
- Sadness - Passive Control (No Intervention): Participants view sadness-related scenario but do not receive any emotion regulation training or distraction tasks. This arm serves as a baseline to measure natural emotional change over time.
- Anxiety - Reconstrual (Experimental): Participants are trained in reconstrual to reinterpret and reduce the perceived threat or negative appraisal of the situation and exposed to anxiety-inducing scenario. The online training includes practice vignette, followed by application of the strategy to the scenario.
  Interventions: Behavioral: Reconstrual Strategy Training
- Anxiety - Repurposing (Experimental): Participants view anxiety-related scenarios and receive training in repurposing, which focuses on changing the goal to alleviate negative feelings. Training and practice exercises are provided online through Qualtrics before applying the strategy to the scenario.
  Interventions: Behavioral: Repurposing Strategy Training
- Anxiety - Active Control (Active Comparator): Participants are presented with anxiety-related scenario followed by a writing distraction task designed to divert attention from negative emotions. This arm controls for the effect of engaging in an active cognitive task unrelated to emotion regulation.
  Interventions: Behavioral: Active Control
- Anxiety - Passive Control (No Intervention): Participants view anxiety-related scenario but do not receive any emotion regulation training or distraction tasks. This arm serves as a baseline to measure natural emotional change over time.

INTERVENTIONS:
Behavioral: Reconstrual Strategy Training — Participants receive training in the reconstrual strategy, which involves recognizing and reinterpreting initial negative appraisals of emotionally challenging situations. The training guides participants to:
  Identify the situation and their initial negative interpretation.
  Generate alternative, balanced explanations that reduce negative emotional impact.
  The goal is to help participants view events from a different, realistic perspective to decrease negative emotions by modifying how they interpret situations.
  Arms: Anxiety - Reconstrual; Sadness - Reconstrual
Behavioral: Repurposing Strategy Training — Participants receive training in the repurposing strategy, which involves adjusting or replacing personal goals to better align with the current situation. The training guides participants to:
  Identify the situation and the original goal that was not met.
  Develop alternative, realistic goals or modify existing ones to reduce the emotional impact of unmet expectations.
  This approach helps participants manage negative emotions by creating meaningful, adaptable goals that fit the reality of the situation.
  Arms: Anxiety - Repurposing; Sadness - Repurposing
Behavioral: Active Control — Participants are asked to carefully copy a neutral descriptive passage without making any changes, focusing solely on transcription accuracy. This task serves as an active control by engaging participants in a cognitive task that requires attention and effort, but does not involve emotion regulation strategies. The task controls for the effects of engagement and time spent on a task without influencing participants' emotional processing.
  Arms: Anxiety - Active Control; Sadness - Active Control

SUMMARY:
The goal of this clinical trial is to learn which reappraisal strategy works better to reduce sadness and anxiety in emerging adults. The main questions it aims to answer are:

What is the effect of emotion regulation strategies (reconstrual, repurposing) on short term negative emotions (anxiety, sadness)?

Does the effectiveness of these strategies vary depending on the type of emotion (anxiety vs. sadness)?

Are reconstrual and repurposing more effective compared to active and passive control conditions?

What is the effect of these strategies on short-term positive emotions (e.g., hope, happiness)?

Researchers will compare reconstrual and repurposing strategies to see which one is more effective in improving emotional outcomes.

Participants will:

be randomly assigned to one of eight conditions in a 4 (Regulation Strategy: Reconstrual, Repurposing, Active Control, Passive Control) × 2 (Emotion Type: Sadness vs. Anxiety) factorial design.

Complete online tasks and surveys about their emotions

DETAILED DESCRIPTION:
This study evaluates the effectiveness of two cognitive reappraisal strategies-reconstrual (reinterpreting the meaning of an event) and repurposing (modifying the personal goal related to the event)-in reducing negative affect and enhancing positive affect in response to emotion-evoking scenarios in emerging adults.

Participants (at least N = 240) will be randomly assigned to one of eight groups in a 2 (Emotion: Sadness vs. Anxiety) × 4 (Strategy: Reconstrual, Repurposing, Active Control, Passive Control) between-subjects factorial design. Each participant will complete standardized emotional induction tasks via written scenarios, followed by their assigned intervention.

Hypotheses

H1: Negative emotions (sadness or anxiety) will significantly decrease following the intervention in the reconstrual and repurposing groups compared to the active and passive control groups. (Main effect of strategy on negative affect)

H2: Positive emotions will increase more in the reconstrual and repurposing groups compared to the passive control group. (Main effect of strategy on positive affect)

H3 (Exploratory): The effectiveness of reconstrual and repurposing strategies may vary by emotion type:

Repurposing may be more effective in sadness scenarios.

Reconstrual may be more effective in anxiety scenarios. (Emotion Type × Strategy interaction)

H4: No significant emotional change is expected in the passive control group. (No time effect)

Study Design

Design Type: Experimental, between-subjects factorial design Design Structure: 2 (Emotion Type: Sadness vs. Anxiety) × 4 (Strategy Condition: Reconstrual, Repurposing, Active Control, Passive Control) Participants: Minimum N = 240 (n = 30 per group), emerging adults (ages ~18-30) Randomization: Random assignment to 1 of 8 groups Blinding: Participants are blind to condition purpose Type of Analysis: Mixed ANOVA

Within-Subject Factor: Time (Post-Scenario vs. Post-Intervention) Between-Subject Factors: Emotion Type × Strategy Group Dependent Variables: Emotional ratings post-intervention (Negative affect (VAS/SAM: anxiety, sadness); Positive affect (VAS/SAM).

Study Flow

1. Initial Assessment Demographics: Only name and age Baseline measures: Scale for contextual reappraisal (SCORE; for trait-level reconstrual and repurposing), GAD-7, PHQ-9
2. Neutral Stimulus A standardized neutral video from Samson et al. (2016) study.
3. Baseline Emotion Assesments: Self-Assessment Manikin (SAM), Visual Analogue Scale (VAS)
4. Random Group Assignment

   Participants randomly assigned to one of eight groups (n=30 per group):

   Sadness - Reconstrual

   Sadness - Repurposing

   Sadness - Active Control

   Sadness - Passive Control

   Anxiety - Reconstrual

   Anxiety - Repurposing

   Anxiety - Active Control

   Anxiety - Passive Control
5. Training Phase Strategy-specific training with a minimum 90-second reading time enforced

   Practice vignette with 30-second enforced reading and comprehension check

   Correct answers allow progression; incorrect answers trigger explanation and acknowledgment before continuing

   Participants rate prior use of the trained strategy in daily life
6. Scenario Exposure Participants read and imagine a standardized written scenario (sadness or anxiety) matched for intensity and controllability (based on pilot data)

40-second enforced reading time

7. Self-Assessment and Rating VAS and SAM administered

Ratings of scenario imaginability and controllability (0-100 scale)

Participants write their first negative thoughts when imagining the scenario

8. Application Phase Participants apply assigned emotion regulation strategy with 90-second minimum enforced duration

Written brief explanation of alternative thoughts used

Post-application ratings with VAS and SAM

Participants rate effectiveness and belief in their reappraisal thoughts (0-100 scale)

9. Manipulation Check In the form of two multiple-choice questions: Participants will be asked to select the instruction that best matched the guideline they received at the beginning of the experiment and to identify the general topic of the scenario they had visualized.

10. Demographics: Exclusion criteria related questions 11. Debriefing Participants view debriefing statement

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Fluent in Turkish
* No current psychiatric treatment or diagnosis (self-reported)
* Willingness to participate and provide informed consent

Exclusion Criteria:

* History of severe psychiatric or neurological disorders
* Current substance use disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Negative Affect | Immediately after vignette exposure vs. immediately after intervention
  (VAS; scale 0-100)
  Participants rate how intensely they feel a target negative emotion (sadness or anxiety) using a Visual Analogue Scale (VAS) from 0 ("Not at all") to 100 ("Extremely").
  Assessment Points:
  Time 1: After reading the emotionally evocative vignette (baseline).
  Time 2: After completing the assigned emotion regulation strategy (post-intervention)
Change in valence and arousal | Immediately after vignette exposure vs. immediately after intervention
  Self-Assessment Manikin (SAM) ratings [Time Frame: Before vs. after intervention]
  A nonverbal pictorial measure of emotional response that assesses two dimensions:
  Valence (pleasant-unpleasant)
  Arousal (high-low) on a 1-9 scale

SECONDARY OUTCOMES:
Change in Positive Affect | Immediately after vignette exposure vs. immediately after intervention
  (VAS; scale 0-100)
PHQ-9 (Patient Health Questionnaire) | Baseline
  Description: A 9-item measure of depressive symptoms over the past two weeks.
  Scoring: 0-27 total score
  Cutoffs:
  5 = mild 10 = moderate 15 = moderately severe 20 = severe
  Use: may explain individual differences in affective response or strategy preference.
GAD-7 (Generalized Anxiety Disorder Scale) | Baseline
  Description: A 7-item scale assessing anxiety symptoms over the past two weeks.
  Scoring: 0 (not at all) to 3 (nearly every day); total score range: 0-21
  Cutoffs:
  5 = mild 10 = moderate 15 = severe
  Assessment Point: baseline
  Use: As a moderator variable to assess if baseline anxiety affects strategy effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ALTAN-ATALAY, Assoc. Prof. Dr, Principal Investigator — Kadir Has University; Burcu UYSAL, Assoc. Prof. Dr, Principal Investigator — Ibn Haldun University
Locations (1):
- Ibn Haldun University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data will be shared upon reasonable request after publication, following approval from the ethics committee and under a data use agreement.

REFERENCES:
- [Background] Samson AC, Kreibig SD, Soderstrom B, Wade AA, Gross JJ. Eliciting positive, negative and mixed emotional states: A film library for affective scientists. Cogn Emot. 2016 Aug;30(5):827-56. doi: 10.1080/02699931.2015.1031089. Epub 2015 May 1. PMID 25929696
- [Background] Kam JWY, Wan-Sai-Cheong L, Zuk AAO, Mehta A, Dixon ML, Gross JJ. A brief reappraisal intervention leads to durable affective benefits. Emotion. 2024 Oct;24(7):1676-1688. doi: 10.1037/emo0001391. Epub 2024 Jun 20. PMID 38900559
- [Background] Uusberg A, Yih J, Taxer JL, Christ NM, Toms T, Uusberg H, Gross JJ. Appraisal shifts during reappraisal. Emotion. 2023 Oct;23(7):1985-2001. doi: 10.1037/emo0001202. Epub 2023 Feb 6. PMID 36745065
- [Background] Wang K, Goldenberg A, Dorison CA, Miller JK, Uusberg A, Lerner JS, Gross JJ, Agesin BB, Bernardo M, Campos O, Eudave L, Grzech K, Ozery DH, Jackson EA, Garcia EOL, Drexler SM, Jurkovic AP, Rana K, Wilson JP, Antoniadi M, Desai K, Gialitaki Z, Kushnir E, Nadif K, Bravo ON, Nauman R, Oosterlinck M, Pantazi M, Pilecka N, Szabelska A, van Steenkiste IMM, Filip K, Bozdoc AI, Marcu GM, Agadullina E, Adamkovic M, Roczniewska M, Reyna C, Kassianos AP, Westerlund M, Ahlgren L, Pontinen S, Adetula GA, Dursun P, Arinze AI, Arinze NC, Ogbonnaya CE, Ndukaihe ILG, Dalgar I, Akkas H, Macapagal PM, Lewis S, Metin-Orta I, Foroni F, Willis M, Santos AC, Mokady A, Reggev N, Kurfali MA, Vasilev MR, Nock NL, Parzuchowski M, Espinoza Barria MF, Vranka M, Kohlova MB, Ropovik I, Harutyunyan M, Wang C, Yao E, Becker M, Manunta E, Kaminski G, Boudesseu J, Marko D, Evans K, Lewis DMG, Findor A, Landry AT, Aruta JJB, Ortiz MS, Vally Z, Pronizius E, Voracek M, Lamm C, Grinberg M, Li R, Valentova JV, Mioni G, Cellini N, Chen SC, Zickfeld J, Moon K, Azab H, Levy N, Karababa A, Beaudry JL, Boucher L, Collins WM, Todsen AL, van Schie K, Vintr J, Bavolar J, Kaliska L, Krizanic V, Samojlenko L, Pourafshari R, Geiger SJ, Beitner J, Warmelink L, Ross RM, Stephen ID, Hostler TJ, Azouaghe S, McCarthy R, Szala A, Grano C, Solorzano CS, Anjum G, Jimenez-Leal W, Bradford M, Perez LC, Cruz Vasquez JE, Galindo-Caballero OJ, Vargas-Nieto JC, Kacha O, Arvanitis A, Xiao Q, Carcamo R, Zorjan S, Tajchman Z, Vilares I, Pavlacic JM, Kunst JR, Tamnes CK, von Bastian CC, Atari M, Sharifian M, Hricova M, Kacmar P, Schrotter J, Rahal RM, Cohen N, FatahModares S, Zrimsek M, Zakharov I, Koehn MA, Esteban-Serna C, Calin-Jageman RJ, Krafnick AJ, Strukelj E, Isager PM, Urban J, Silva JR, Martoncik M, Ocovaj SB, Sakan D, Kuzminska AO, Djordjevic JM, Almeida IAT, Ferreira A, Lazarevic LB, Manley H, Ricaurte DZ, Monteiro RP, Etabari Z, Musser E, Dunleavy D, Chou W, Godbersen H, Ruiz-Fernandez S, Reeck C, Batres C, Kirgizova K, Muminov A, Azevedo F, Alvarez DS, Butt MM, Lee JM, Chen Z, Verbruggen F, Ziano I, Tumer M, Charyate ACA, Dubrov D, Tejada Rivera MDCMC, Aberson C, Palfi B, Maldonado MA, Hubena B, Sacakli A, Ceary CD, Richard KL, Singer G, Perillo JT, Ballantyne T, Cyrus-Lai W, Fedotov M, Du H, Wielgus M, Pit IL, Hruska M, Sousa D, Aczel B, Hajdu N, Szaszi B, Adamus S, Barzykowski K, Micheli L, Schmidt ND, Zsido AN, Paruzel-Czachura M, Muda R, Bialek M, Kowal M, Sorokowska A, Misiak M, Mola D, Ortiz MV, Correa PS, Belaus A, Muchembled F, Ribeiro RR, Arriaga P, Oliveira R, Vaughn LA, Szwed P, Kossowska M, Czarnek G, Kielinska J, Antazo B, Betlehem R, Stieger S, Nilsonne G, Simonovic N, Taber J, Gourdon-Kanhukamwe A, Domurat A, Ihaya K, Yamada Y, Urooj A, Gill T, Cadek M, Bylinina L, Messerschmidt J, Kurfali M, Adetula A, Baklanova E, Albayrak-Aydemir N, Kappes HB, Gjoneska B, House T, Jones MV, Berkessel JB, Chopik WJ, Coksan S, Seehuus M, Khaoudi A, Bokkour A, El Arabi KA, Djamai I, Iyer A, Parashar N, Adiguzel A, Kocalar HE, Bundt C, Norton JO, Papadatou-Pastou M, De la Rosa-Gomez A, Ankushev V, Bogatyreva N, Grigoryev D, Ivanov A, Prusova I, Romanova M, Sarieva I, Terskova M, Hristova E, Kadreva VH, Janak A, Schei V, Sverdrup TE, Askelund AD, Pineda LMS, Krupic D, Levitan CA, Johannes N, Ouherrou N, Say N, Sinkolova S, Janjic K, Stojanovska M, Stojanovska D, Khosla M, Thomas AG, Kung FYH, Bijlstra G, Mosannenzadeh F, Balci BB, Reips UD, Baskin E, Ishkhanyan B, Czamanski-Cohen J, Dixson BJW, Moreau D, Sutherland CAM, Chuan-Peng H, Noone C, Flowe H, Anne M, Janssen SMJ, Topor M, Majeed NM, Kunisato Y, Yu K, Daches S, Hartanto A, Vdovic M, Anton-Boicuk L, Forbes PAG, Kamburidis J, Marinova E, Nedelcheva-Datsova M, Rachev NR, Stoyanova A, Schmidt K, Suchow JW, Koptjevskaja-Tamm M, Jernsather T, Olofsson JK, Bialobrzeska O, Marszalek M, Tatachari S, Afhami R, Law W, Antfolk J, Zuro B, Van Doren N, Soto JA, Searston R, Miranda J, Damnjanovic K, Yeung SK, Krupic D, Hoyer K, Jaeger B, Ren D, Pfuhl G, Klevjer K, Corral-Frias NS, Frias-Armenta M, Lucas MY, Torres AO, Toro M, Delgado LGJ, Vega D, Solas SA, Vilar R, Massoni S, Frizzo T, Bran A, Vaidis DC, Vieira L, Paris B, Capizzi M, Coelho GLH, Greenburgh A, Whitt CM, Tullett AM, Du X, Volz L, Bosma MJ, Karaarslan C, Sarioguz E, Allred TB, Korbmacher M, Colloff MF, Lima TJS, Ribeiro MFF, Verharen JPH, Karekla M, Karashiali C, Sunami N, Jaremka LM, Storage D, Habib S, Studzinska A, Hanel PHP, Holford DL, Sirota M, Wolfe K, Chiu F, Theodoropoulou A, Ahn ER, Lin Y, Westgate EC, Brohmer H, Hofer G, Dujols O, Vezirian K, Feldman G, Travaglino GA, Ahmed A, Li M, Bosch J, Torunsky N, Bai H, Manavalan M, Song X, Walczak RB, Zdybek P, Friedemann M, Rosa AD, Kozma L, Alves SG, Lins S, Pinto IR, Correia RC, Babincak P, Banik G, Rojas-Berscia LM, Varella MAC, Uttley J, Beshears JE, Thommesen KK, Behzadnia B, Geniole SN, Silan MA, Maturan PLG, Vilsmeier JK, Tran US, Izquierdo SM, Mensink MC, Sorokowski P, Groyecka-Bernard A, Radtke T, Adoric VC, Carpentier J, Ozdogru AA, Joy-Gaba JA, Hedgebeth MV, Ishii T, Wichman AL, Roer JP, Ostermann T, Davis WE, Suter L, Papachristopoulos K, Zabel C, Onie S, Ebersole CR, Chartier CR, Mallik PR, Urry HL, Buchanan EM, Coles NA, Primbs MA, Basnight-Brown DM, IJzerman H, Forscher PS, Moshontz H. A multi-country test of brief reappraisal interventions on emotions during the COVID-19 pandemic. Nat Hum Behav. 2021 Aug;5(8):1089-1110. doi: 10.1038/s41562-021-01173-x. Epub 2021 Aug 2. PMID 34341554
- [Background] Uusberg A, Ford B, Uusberg H, Gross JJ. Reappraising reappraisal: an expanded view. Cogn Emot. 2023 May-Jun;37(3):357-370. doi: 10.1080/02699931.2023.2208340. Epub 2023 May 10. PMID 37161355
- [Background] Aldao A. The Future of Emotion Regulation Research: Capturing Context. Perspect Psychol Sci. 2013 Mar;8(2):155-72. doi: 10.1177/1745691612459518. PMID 26172497